CLINICAL TRIAL: NCT07029100
Title: Feasibility of ORGAnoids in Routine Clinical Practice for Molecular Analysis of the GLIOvascular Niche in Patients With Primary Brain Tumors.
Acronym: ORGA-GLIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHB24.05; 2024-A02153-44 (Other: ANSM)
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: glioblastoma; organoide; molecular analysis
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex-vivo Organoid culture (Experimental): ex-vivo organoid culture after tumor resection
  Interventions: Other: Ex-vivo organoid culture

INTERVENTIONS:
Other: Ex-vivo organoid culture — ex-vivo organoid cultures composed of tumor cells within their microenvironment (glioblastoma organoid - GBO) and intra- and peri-tumoral blood vessels (blood vessel organoid - BVO), derived from perioperative samples obtained during complete or partial surgical resection

SUMMARY:
The main goal of ORGA-GLIO trial is to establish the feasibility in routine clinical practice of ex-vivo organoid cultures composed of tumor cells within their microenvironment (glioblastoma organoid - GBO) and intra- and peri-tumoral blood vessels (blood vessel organoid - BVO), derived from perioperative samples obtained during complete or partial surgical resection in patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
The ORGA-GLIO study will be conducted in two stages:

First stage: Establishment of the clinical-biological collection and addressing the primary objective.

Step 1: Generation of tumor organoids (Glioblastoma Organoids - GBO), vascular organoids (Blood Vessel Organoids - BVO), and cell lines.

Step 2: Phenotypic and molecular analyses of tumor and vascular organoids up to 7 days.

Second stage: Utilization of the biological collection of organoids and blood samples.

Utilization of the organoid collection and investigation of associations between the molecular and phenotypic and clinical and survival data collected during patient follow-up visits.

Correlation of organoid evolution under experimental treatment procedure and evolution of plasma-based biomarker from corresponding patients and along first-line treatment schedule.

All patients will be planned to receive standard of care for glioblastoma after resection, namely radiotherapy+temozolomide and TTFields.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, adult (age ≥ 18 years),
* Suspected of having a high-grade glioma based on preoperative multimodal MRI,
* With an indication for tumor resection surgery,
* And in a clinical condition suitable to undergo adjuvant treatment consisting of radiotherapy (normo- or hypo-fractionated) combined with temozolomide, with or without low-frequency electric fields (Tumor-Treating Fields®).

Exclusion Criteria:

* Current tumor pathology or history of tumor pathology in remission for less than 2 years
* Pregnant or breastfeeding women,
* Patients unable to understand the study for any reason or unable to comply with trial requirements (language barriers, psychological or geographical issues, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Ex-vivo organoid culture feasability | 7 days
  Proportion (in number of patients) of phenotypically and molecularly exploitable tumor and vascular organoid models (GBO+BVO) seven days after diagnostic neurosurgical removal (complete or partial excision) in patients with glioblastoma

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Groupe Hospitalier du Havre, Le Havre
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No